CLINICAL TRIAL: NCT06017401
Title: Comparison of The Effect of Oblique Subcostal Transversus Abdominis Plane Block and Transmuscular Quadratus Lumborum Block on Postoperative Analgesia and Quality of Recovery in Patients Undergoing Laparoscopic Gynecological Surgery
Brief Title: Oblique Subcostal Transversus Abdominis Plane Block Versus Transmuscular Quadratus Lumborum Block for Pain Management in Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Kübra Cebeci, Research Assistant, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UludagU-KCebeci-001
Record Dates: First submitted 2023-08-20; First posted 2023-08-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain; Surgery
Keywords: Postoperative pain; Pain management; Oblique subcostal transversus abdominis plane block; Transmuscular quadratus lumborum block; Quality of Recovery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group OSTAP (Active Comparator): The investigator will perform oblique subcostal transversus abdominis plane block to that patient group for postoperative analgesia
  Interventions: Procedure: Oblique Subcostal Transversus Abdominis Plane Block
- Group TQLB (Active Comparator): The investigator will perform transmuscular quadratus lumborum block to that patient group for postoperative analgesia
  Interventions: Procedure: Transmuscular Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Oblique Subcostal Transversus Abdominis Plane Block — The investigator will perform oblique subcostal transversus abdominis plane block to that patient group for postoperative analgesia
  Arms: Group OSTAP
Procedure: Transmuscular Quadratus Lumborum Block — The investigator will perform transmuscular quadratus lumborum block to that patient group for postoperative analgesia
  Arms: Group TQLB

SUMMARY:
Laparoscopic gynecological surgery causes postoperative pain.The primary objective of this study is to compare the effect of ultrasound (US)-guided oblique subcostal transversus abdominis plane block (OSTAP) on 24-hour total analgesic consumption with transmuscular quadratus lumborum block (TQLB).

DETAILED DESCRIPTION:
Patients between the ages of 18-65, who will undergo laparoscopic gynecological surgery, American Society of Anesthesiologists (ASA) class I-II-III, Body Mass Index (BMI) in the range of 18-25 kg/m², and who will use 3 or 4 trocar for surgery will be included in the study. Patients will be randomized into two groups. OSTAP block will be performed for OSTAPB group and TQL block will be performed for TQLB group. Patients will be administered postoperative 4x500 mg iv paracetamol as needed (if Visual Analogue Scale (VAS) score is 4 or higher). If the VAS score remains at 4 or higher 30 minutes after paracetamol administration, 1 mg/kg iv tramadol will be administered as a rescue analgesic (with a daily maximum dose of 400 mg). The primary outcome is to compare the total analgesic consumption within the first 24 hours after surgery. The secondary outcome is to compare the time to the first postoperative analgesic requirement, VAS scores at rest and on movement, and assess the impact of these two blocks on the quality of recovery using the QOR-15 scale

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65
* Patients who will undergo laparoscopic gynecological surgery
* ASA I-II-III patients
* Body Mass Index (BMI) in the range of 18-25 kg/m²
* Patients who will undergo surgery using 3 or 4 trocars

Exclusion Criteria:

* ASA IV-V
* Patients with a known or suspected allergy to local anesthetics
* Coagulopathy
* Injection site infection
* Severe neurological or psychiatric disorders
* Severe cardiovascular disease
* Liver failure
* Kidney failure (glomerular filtration rate <15 ml/min/m²)
* Chronic opioid use (>6 months)
* Surgical durations less than 45 minutes or greater than 120 minutes

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Postoperative 24 hours total analgesic consumption | 24 hours postoperatively
  The primary outcome is to compare the total consumption of paracetamol and tramadol within the first 24 hours after surgery.

SECONDARY OUTCOMES:
The time to the first analgesic requirement, VAS scores and QOR-15 scores of the patients | 24 hours postoperatively
  The secondary outcomes are to compare the time to the first postoperative analgesic requirement, VAS scores at 0, 30th min and 1, 2, 6, 12, 18, 24th hours at rest and on movement, and assess the impact of these two blocks on the quality of recovery using the QoR-15 scale.
  A visual analogue scale (VAS) requires the patient to rate their pain on a scale of 0-10, where 0 represents no pain and 10 represents the worst pain imaginable.
  The QoR-15 scale is a unidimensional measurement of quality of recovery measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Faculty of Medicine, Bursa, Turkey (Türkiye)